CLINICAL TRIAL: NCT05388162
Title: Smart-phone Based Cervical Imaging Device Compared With a Standard Culposcope for the Detection of Cervical Dysplasia A Non-inferiority Evaluation.
Brief Title: A Non-inferiority Evaluation of a Smart-phone Based Cervical Imaging Device.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Bruce Kahn, PI, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Smart-phone based culposcope
Record Dates: First submitted 2015-11-27; First posted 2022-05-24 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer screening,colposcopy,smartphone
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- coposcopy (Other): patients undergoing colposcopy will have images taken of the cervix with a standard colposcope and the Mobile colposcope. de-identified images from both devices will then be entered into a custom colposcopic image evaluation program. Images will then be randomly evaluated by expert colposcopists as normal, abnormal or cannot evaluate. On abnormal images, the most abnormal point on the images will be marked as teh recommended biopsy site. Scoring for images from the standard colposcope will be compared with that for the Mobile Colposcope.
  Interventions: Device: Mobile colposcope

INTERVENTIONS:
Device: Mobile colposcope — It is a comparison trial - Comparing a standard colposcpoe with a smart-phone based colpsocpe.

SUMMARY:
When a woman has an abnormal pap smear or tests positive for a high risk strain of the HPV virus, the current standard of care includes culposcopic examination of the cervix with biopsy. A culposcope is essentially a microscope for examining the cervix. Culposcopes cost $5-10,000 each. The device being tested in this trial is an adaptor for a smart phone that will cost ~ $125. The larger goal of this line of studies see if the images obtained using the smart phone adaptor are non-inferior to those obtained with standard culposcopes. If the device is found to provide images equal to those of standard culposscopes, it could save thousands of dollars in healthcare expenditure currently that go to the purchase and maintenance of culposcopes. This has potential world-wide applications, especially for resource poor countries. This initial trial is a non-inferiority trial to compare the images obtained with the smart phone based device of those obtained by a standard culposcope

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria: adult women with abnormal pap smear or HPV virus testing referred for culposcopy -

Exclusion Criteria: none

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Determine of the smart-phone based cervical imaging device provides non-inferior image to that obtained using a standard culposcope for the detecton of cervical dysplasia | 1 day
  See above.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kahn, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Clinic, San Diego, California, United States